CLINICAL TRIAL: NCT03509649
Title: The Impact of Practitioner and Instructional Set on Subject Expectations of Cervical Spine Manipulation
Brief Title: Impact of Practitioner and Instructional Set on Subject Perceptions and Expectations of Cervical Spine Manipulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Emilio J Puentedura, PT, DPT, PhD, Principal Investigator, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1144771
Record Dates: First submitted 2018-04-09; First posted 2018-04-26 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants randomly assigned to one of 2 instructional sets (positive/ negative) and randomly assigned to one of 2 practitioner experience levels (experienced/ novice)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experienced - Positive (Experimental): Participants will receive cervical spine manipulation after being given a positive description of the technique from an experienced clinician
  Interventions: Procedure: Cervical spine manipulation
- Experienced - Negative (Experimental): Participants will receive cervical spine manipulation after being given a negative description of the technique from an experienced clinician
  Interventions: Procedure: Cervical spine manipulation
- Novice - Positive (Active Comparator): Participants will receive cervical spine manipulation after being given a positive description of the technique from a novice clinician
  Interventions: Procedure: Cervical spine manipulation
- Novice - Negative (Active Comparator): Participants will receive cervical spine manipulation after being given a negative description of the technique from a novice clinician
  Interventions: Procedure: Cervical spine manipulation

INTERVENTIONS:
Procedure: Cervical spine manipulation — High-velocity low-amplitude thrust joint manipulation to the cervical spine

SUMMARY:
Determine effects of perceptions and expectations on experience of cervical spine manipulation

DETAILED DESCRIPTION:
The purpose of this study is to better understand how therapists may affect a patient's thoughts/ beliefs/ opinions on cervical spine (neck) manipulation. Current evidence suggests that patients who have a positive expectation about neck manipulation are more likely to report benefit from it, and we wish to determine if the perceived experience level of the therapist and the words they use to describe neck manipulation will affect the patient's perception.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years;
2. must report having no current episode of mechanical neck pain;
3. must be willing to participate;
4. must indicate they have not had their neck manipulated by a physical therapist, osteopath or chiropractor within the last 5 years.

Exclusion Criteria:

1. 'Red flag' items indicated in your Neck Medical Screening Questionnaire such as: history of a tumor, bone fracture, metabolic diseases, rheumatoid arthritis, osteoporosis, severe atherosclerosis, prolonged history of steroid use, heart disease, and stroke.
2. History of neck whiplash injury.
3. Diagnosis from your physician of cervical spinal stenosis (narrowing of spinal canal) or presence of symptoms (pain, pins and needles, numbness) in both arms.
4. Presence of central nervous system involvement such as exaggerated reflexes, changes in sensation in the hands or face, muscle wasting in the hands, altered taste, and presence of abnormal reflexes.
5. Evidence of neurological signs suggesting nerve root entrapment (pinched nerve in the neck).
6. Prior surgery to your neck or upper back.
7. A medical condition which may change your sensation of pain or pressure pain thresholds (i.e. taking analgesics, sedatives, history of substance abuse, or cognitive deficiency).
8. Diagnosis from your physician of fibromyalgia syndrome.
9. Currently pregnant, or think you may be pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-05-17 (Estimated); Study Completion 2019-05-17 (Estimated)

PRIMARY OUTCOMES:
Global Perceived Effect Scale (GPE) | Immediate
  7 point Likert scale anchored with "1" completely recovered to "7" worse than ever.

SECONDARY OUTCOMES:
Perception of comfort scale | Immediate
  5 point Likert scale ranging from 1 "very comfortable" to 5 "very uncomfortable
Beliefs about cervical spine manipulation | Immediate
  6 questions determining participant's beliefs about safety, comfort and effectiveness of spinal manipulation. Likert scale with statements participants can 'completely disagree', 'somewhat disagree', 'neutral', 'somewhat agree', or 'completely agree' with

CONTACTS AND LOCATIONS:
Overall Officials: Emilio J Puentedura, DPT, PhD, Principal Investigator — Baylor University
Locations (1):
- University of Nevada Las Vegas - Department of Physical Therapy, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided